CLINICAL TRIAL: NCT06805851
Title: Thermoregulatory Responses to Heat Stress in Adults With Major Depressive Disorder With and Without Antidepressant Treatment
Brief Title: Impact of Depression on Thermoregulation
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, W. Larry Kenney, Professor, Penn State University
Other Study IDs: Study26326
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression; Selective Serotonin Reuptake Inhibitor
Keywords: thermoregulation; heat stress; depression; selective serotonin reuptake inhibitors; serotonin norepinephrine reuptake inhibitors
MeSH Terms: conditions — Depression; Heat Stress Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-depressed
- Depressed: adults with clinically diagnosed major depressive disorder
- SSRI: adults with clinically diagnosed major depressive disorder currently taking a physician prescribed selective serotonin reuptake inhibitor as treatment.
- SNRI: adults with clinically diagnosed major depressive disorder currently taking a physician prescribed serotonin norepinephrine reuptake inhibitor as treatment.

SUMMARY:
The purpose of this study is to determine if, compared to non-depressed adults, differences exist in skin blood flow and sweating responses to passive heat stress in adults with clinically diagnosed depression, those with depression who are prescribed and taking SSRIs and those with depression who are prescribed and taking SNRIs.

DETAILED DESCRIPTION:
Four groups will be recruited to examine the impact of major depressive disorder and pharmaceutical treatments on thermoregulatory heat loss mechanisms. Adults without MDD, adults with MDD, adults with MDD currently prescribed and taking selective serotonin reuptake inhibitors as treatment, and adults with MDD currently prescribed and taking serotonin norepinephrine reuptake inhibitors as treatment will be recruited to completed a passive heat stress experiment. All subjects will sign an informed consent form and undergo a medical screening prior to participation. Each subject will complete 1 passive heat stress experiment in which body temperature will be using a water perfused suit. During passive heating, body temperature, skin blood flow, and local and whole-body sweat rates will be continuously measured and recorded to compare heat stress responses between groups.

ELIGIBILITY:
Inclusion Criteria:

* Non-depressed adults aged 18-40 years;
* OR adults aged 18-40 years with clinically diagnosed major depressive disorder according to DSM-V criteria not currently receiving antidepressant treatment;
* OR adults aged 18-40 years with clinically diagnosed major depressive disorder with at least 2 weeks of treatment with a selective serotonin reuptake inhibitor;
* OR aged 18-40 years adults with clinically diagnosed major depressive disorder with at least 2 weeks of treatment with a serotonin norepinephrine reuptake inhibitor;
* All participants will be asymptomatic and no signs/symptoms of disease according to the American College of Sports Medicine 10th edition Guidelines for Exercise Testing and Prescription (chest pain or pressure, dizziness, joint pain, and signs of cardiovascular disease);
* Systolic blood pressure 140 mmHg and diastolic pressure 90 mmHg at screening;
* Non-diabetic
* Not taking any other medications that might affect the physiological variables of interest (beta blockers, tricyclic antidepressants, antipyretics, diuretics, etc.);;
* Between the 20th and 80th percentiles for sex- and age-appropriate VO2max according to the American College of Sports Medicine 10th edition Guidelines for Exercise Testing and Prescription;
* English proficiency;
* Capable of providing informed consent.

Exclusion Criteria:

* BMI > 35
* Are pregnant or planning to become pregnant in the next 12 months;
* Concurrently participate in another study involving physical activity or weight loss;
* Plan to have surgery or relocate outside the area within the next year;
* Medications that could alter cardiovascular or thermoregulatory responses to exercise (beta blockers, antipyretics, tricyclic antidepressants, diuretics, etc.);
* Allergy to latex or adhesive;
* Tobacco use;
* Illegal/recreational drug use;
* Exertional chest pain or musculoskeletal pain;
* Contraindications to a maximal exercise test or an indication for early termination of the exercise test according to the American College of Sports Medicine 10th edition Guidelines for Exercise Testing and Prescription;
* Abnormal resting or exercise electrocardiogram (ECG);
* Any bleeding disorders, gastric ulcers, allergies to NSAIDS, asthma, kidney/liver disorders, and taking any other anticoagulants;
* History of Crohn's disease, diverticulitis, or similar gastrointestinal disease;
* Co-morbid psychiatric disorders (psychosis, schizophrenia, bipolar disorder, panic disorder, obsessive compulsive disorder, etc.);
* Active suicidal ideation (moderate or high suicidality);
* Use of psychoactive or psychopharmacological drugs other than SSRI and SNRIs within one year of participating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from Centre County Pennsylvania including on the Penn State University campus.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow | Monitored continuously during the passive heating experimental trial, about 2 hours.
  Skin blood flow response to whole body heating is continuously monitored during the experimental trial, about 2 hours.
Local Sweat Rate | Monitored continuously during the passive heating experimental trial, about 2 hours.
  A small sweat capsule is placed on the forearm for the duration of the passive whole body heating experiment, about 2 hours.
Core Temperature | Monitored continuously during the passive heating experimental trial, about 2 hours.
  Changes in body temperature are measured through a telemetry pill swallowed before each experiment.

SECONDARY OUTCOMES:
Body Mass | Will be measured once immediately before and once immediately after the passive heating experimental trail.
  Body mass is measured on a scale before and after the passive heating experimental trail.

CONTACTS AND LOCATIONS:
Overall Officials: W. Larry Kenney, Principal Investigator — The Pennsylvania State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No